CLINICAL TRIAL: NCT00291785
Title: Phase I/II Study of CT-2106 in Combination With Infusional 5-fluorouracil/Folinic Acid (5-FU/FA)(de Gramont Schedule) as Second Line in Patients With Metastatic Colorectal Cancer Failing an Oxaliplatin Plus 5-FU/FA Regimen
Brief Title: Phase I/II CT 2106 and 5-FU/FA in Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Igor Gorbatchevsky,M.D., Cell Therapeutics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM201
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; camptothecin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — polyglutamate camptothecin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CT-2106 — CT-2106 as 10 minute infusion on days 1, 15 & 29 of each 42-day cycle
Drug: Folinic acid — Folinic acid 200 mg IV 1 hour after CT-2106 infusion on days 1, 2, 15, 16, 29 and 30
Drug: 5-FU (fluorouracil) — 5-FU following CT-2106 and folinic acid infusions @ 400 mg/m² IV bolus then 5-FU 600 mg/m² as a 22 hour IV infusion on Days 1, 2, 15, 16, 29, and 30.

SUMMARY:
CT-2106, a camptothecin (CPT) conjugate, is a new generation of topoisomerase I inhibitors designed to deliver higher, more effective chemotherapy to tumor tissue with less toxicity to normal tissues. The objective of this study is to determine the dose limiting toxicities, safety profile and antitumor activity of CT-2016 in combination with 5-FU and folic acid for the treatment of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic colorectal adenocarcinoma, failing one prior treatment containing oxaliplatin plus 5-FU/FA
* At least one measurable lesion according to RECIST criteria for both Phase I and II
* ECOG performance status 0 or 1
* Adequate hematologic, renal and hepatic function
* Wash out period of at least 4 weeks from surgery, 4 weeks from radiotherapy

Exclusion Criteria:

* Past or concurrent history of neoplasm other than colorectal adenocarcinoma, except curatively treated non melanoma skin cancer or in situ carcinoma of the cervix.
* Pregnant or lactating patients
* Prior treatment with camptothecins
* Presence or history of CNS metastasis or carcinomatous leptomeningitis
* Current active infection per investigator assessment
* Unresolved bowel obstruction or partial obstruction, uncontrolled Crohn's disease or ulcerative colitis
* Current history of chronic diarrhea greater than or equal to grade 1 (CTCAE version 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-01; Primary Completion 2007-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Phase I: determine the Maximum Tolerated Dose, dose limiting toxicities, safety profile and antitumor activity | Each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Barone C., M.D., Principal Investigator — Policlinico Universitario "A.Gemelli"
Locations (2):
- Italy (2):
  - Policlinico Universitario "A.Gemelli", Rome
  - Istituto Clinico Humanitas, Rozzano